CLINICAL TRIAL: NCT02792010
Title: Feasibility and Reproducibility of T1 Rho MRI in the Evaluation of Hip Cartilage
Acronym: CARHAT02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL14_0235
Record Dates: First submitted 2016-05-26; First posted 2016-06-07 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
Keywords: T1rho MRI; hip; cartilage; Healthy participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- T1rho MRI (Experimental): Patients included had hip cartilage MRI with acquisition of T1rho MRI sequence.
  Interventions: Device: Hip cartilage MRI

INTERVENTIONS:
Device: Hip cartilage MRI — Hip cartilage MRI

SUMMARY:
Hip osteoarthritis is a frequent and invalidating disease. Early detection of cartilage modifications could provide better patient treatment. The T1rho MRI sequence allows the quantification of the cartilage signal that is correlated to modifications of the cartilage matrix, notably of the proteoglycans. The primary objective is to evaluate normal values of hip cartilage in vivo using T1rho MRI in healthy subjects and the reproducibility of the measurements. T1rho and T2 mapping sequences were acquired twice during the same session with 30 minutes interval to see if values were modified after a 30 minutes delay in a supine position. The secondary objective was to assess the correlation between T1rho and T2 values.

ELIGIBILITY:
Inclusion Criteria:

* BMI <30
* Accepting to participate in the study and signed the written informed consent
* Covered by a health insurance system

Exclusion Criteria:

* Pregnant woman or risk of pregnancy
* MRI contraindication
* Protected adults
* Language barrier
* Previous or current hip pain

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Quantification of the cartilage signal at T1rho MRI | Up to one month after inclusion (Visit 1)
  T1rho values of total hip cartilage and for each sub-region (mean, standard deviation, histogram)

SECONDARY OUTCOMES:
Quantification of the cartilage signal at T1rho MRI | 15 (+/- 7) days after visit 1 (Visit 2)
  T1rho values of total hip cartilage and for each sub-region (mean, standard deviation, histogram)
Quantification of the cartilage signal at T2 MRI | Up to one month after inclusion (Visit 1)
  T2 values of total hip cartilage and for each sub-region (mean, standard deviation, histogram)
Quantification of the cartilage signal at T2 MRI | 15 (+/- 7) days after visit 1 (Visit 2)
  T2 values of total hip cartilage and for each sub-region (mean, standard deviation, histogram)
Presence of cartilage lesions | Up to one month after inclusion (Visit 1)
  Morphological sequence to determine focal lesions
Presence of cartilage lesions | 15 (+/- 7) days after visit 1 (Visit 2)
  Morphological sequence to determine focal lesions

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste PIALAT, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon - Hôpital Edouard Herriot Pavillon B Radiologie, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nemeth A, Di Marco L, Boutitie F, Sdika M, Grenier D, Rabilloud M, Beuf O, Pialat JB. Reproducibility of in vivo magnetic resonance imaging T1 rho and T2 relaxation time measurements of hip cartilage at 3.0T in healthy volunteers. J Magn Reson Imaging. 2018 Apr;47(4):1022-1033. doi: 10.1002/jmri.25799. Epub 2017 Jun 26. PMID 28650110